CLINICAL TRIAL: NCT06938945
Title: Remote Symptom Monitoring on Patient-Reported Outcomes With Nudge Strategies Among Patients With Tumor in China: A Randomized Controlled Trial
Brief Title: Remote Symptom Monitoring on Patient-Reported Outcomes With Nudge Strategies Among Patients With Tumor in China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wei Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Wei Xiaoping, PhD Candidate,China Center for Health Development Studies, Peking University, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00001052-24066
Record Dates: First submitted 2025-03-25; First posted 2025-04-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: receive PRO（patient reported outcomes） interventions (Experimental)
  Interventions: Behavioral: Digitized patient-reported outcomes
- Control Group：usual care (not receive PRO intervention) (No Intervention)

INTERVENTIONS:
Behavioral: Digitized patient-reported outcomes — Patients fill out the PRO scale regularly online through a specific cell phone program or website, which intelligently analyzes the patient's physical condition, gives symptom management recommendations (which are based on clinical guidelines and expert consensus, and are updated monthly by oncology clinical experts during the study period), and sends alerts to clinical caregivers when the scale scores are abnormal.
  Arms: Intervention Group: receive PRO（patient reported outcomes） interventions

SUMMARY:
The goal of this clinical trial is to design a digital PRO intervention model applicable to patients with hepatocellular carcinoma, and The main questions it aims to answer are:

* Can symptom management through patients' regular completion of the PRO scale promote self-understanding, self-management and timely seeking of medical help, enable healthcare professionals to accurately and efficiently understand how patients really feel and respond in a timely manner, and ultimately improve health outcomes?
* Can digital interventions significantly improve outcomes such as symptom control and quality of life in cancer patients? Researchers divided participants into an intervention group and a control group and compared them to see if digital interventions could improve patient health outcomes.

Participants will:

* Subjects in the intervention group will be asked to report symptom information weekly (7-day natural week, hereafter) via the public number, and the back office will give symptom management advice or issue alerts based on the filling. Control subjects will not receive PRO intervention.
* Participants can offer to withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

1. The patients are aged between 18 and 75 years old;
2. The patients have been diagnosed with locally advanced or metastatic liver cancer through pathological or imaging examinations;
3. The patients are currently receiving or have completed PD-1 monotherapy or PD-1 combination therapy;
4. The patients can participate in this study as per the requirements of the research protocol;
5. The patients voluntarily sign the informed consent form.

Exclusion Criteria:

1. The patients have cognitive impairment or are unable to clearly identify their own symptoms and feelings;
2. The patients are illiterate or unable to understand the research content for other reasons;
3. The patients are currently participating in other clinical trials that may affect this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-05-24 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Health-Related quality of life | 6 months
  EORTC QLQ-C30 Quality of Life Scale(European Organization for Research and Treatment of Cancer Quality of Life Questionnaire) The EORTC QLQ-C30 (Version 3) uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 (Version 3) uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.

SECONDARY OUTCOMES:
Change in patient-reported hepatocellular carcinoma symptoms | 6 months
  PRO questionnaire
Mental health | 6 months
  PHQ-9 Scale((Patient Health Questionnaire-9) The total score can range from 0 to 27. Higher scores indicate greater severity of depression.
Survival period | 6 months
Treatment satisfaction | 6 months
  PRO questionnaire
Treatment compliance | 6 months
  The Morisky Medication Adherence Scale (MMAS-8) The total score of the MMAS-8 scale is the sum of the scores of 8 questions. The score range is 0 to 8 points. The higher the score, the better the medication compliance. A score of 8 indicates good compliance; A score of 6 to 7 indicates moderate compliance. A score less than 6 indicates poor compliance.
The number of times the official account functions are used | 6 months
  The native statistics system of the WeChat Official Account backend
The number of visits to the outpatient department, inpatient department and emergency department | 6 months
  PRO questionnaire
Direct medical costs | 6 months
Direct non-medical costs | 6 months
Indirect cost | 6 months
Health State Utility | 6 months
  EuroQol 5-Dimension 5-Level (EQ-5D-5L) The scale measures quality of life on a 5-component scale.For each dimension, based on the level selected by the respondents, the score for that level is given respectively, with the highest being 5 points and the lowest being 1 point. Then add up the scores of all dimensions to obtain the score of the entire rating scale, with a maximum of 25 points and a minimum of 5 points.The higher the score, the lower the health state utility.

CONTACTS AND LOCATIONS:
Locations (1):
- China Center for Health Development Studies, Peking University, Haidian, Beijing Municipality, China